CLINICAL TRIAL: NCT06555315
Title: Pilot Non-inferiority Study Investigating Daily Versus Every Other Day Dosing of Oral Iron in Premature Infants.
Brief Title: Pilot Trial Investigating Every Other Day Dosing of Oral Iron in Premature Infants (IQONic)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHRISTUS Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-091
Record Dates: First submitted 2024-07-31; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Very Low Birth Weight Infant; Premature Infants; Anemia of Prematurity; Iron Deficiency, Anaemia in Children; Extremely Low Birth Weight
Keywords: Premature infants; Iron; anemia of prematurity; iron deficiency
MeSH Terms: conditions — Premature Birth; Anemia; Iron Deficiencies | interventions — Iron

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A statistician who is blinded to the study allocation will analyze the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): After the infant achieves full enteral feeds, the infant is started on 6 mg/kg of oral iron daily supplementation. The dose of 6 mg/kg of enteral iron was chosen based on the aforementioned recommendations with evidence of its safety, while minimizing the need to increase the enteral iron dosage if an infant were to be started on ESAs where a dose of 6 mg/kg of enteral iron supplementation is the standard practice. Phlebotomy to obtain a complete blood count, reticulocyte count, and reticulocyte hemoglobin count is pursued the Monday after starting iron supplementation and every 2 weeks thereafter to weeks to monitor hematocrit or hemoglobin levels and iron status.
  Interventions: Dietary Supplement: 6 mg/kg of oral iron as ferrous sulfate administered every day.
- Intervention Group (Experimental): After the infant achieves full enteral feeds, the infant is started on 6mg/kg of oral iron supplementation administered every other day. The dose of 6 mg/kg of enteral iron was chosen based on the aforementioned recommendations with evidence of its safety, while minimizing the need to increase the enteral iron dosage if an infant were to be started on ESAs where a dose of 6 mg/kg of enteral iron supplementation is the standard practice. Phlebotomy to obtain a complete blood count, reticulocyte count, and reticulocyte hemoglobin count is pursued the Monday after starting iron supplementation and every 2 weeks thereafter to weeks to monitor hematocrit or hemoglobin levels and iron status.
  Interventions: Dietary Supplement: 6 mg/kg of oral iron as ferrous sulfate administered every other day.

INTERVENTIONS:
Dietary Supplement: 6 mg/kg of oral iron as ferrous sulfate administered every other day. — 6mg/kg of oral iron as ferrous sulfate administered every other day instead of 6 mg/kg of oral iron daily supplementation.
  Arms: Intervention Group
Dietary Supplement: 6 mg/kg of oral iron as ferrous sulfate administered every day. — 6 mg/kg of oral iron as daily ferrous sulfate instead of 6mg/kg of oral iron supplementation administered every other day.
  Arms: Control Group

SUMMARY:
Study focuses on determining if daily versus every-other-day (EOD) oral iron at the same dose per kilogram per day will achieve similar incidence of iron replete status at 36 weeks post-menstrual age in premature neonates

DETAILED DESCRIPTION:
Iron is an important component of hemoglobin, and an essential part of erythropoiesis. It is also a necessary micronutrient for rapidly proliferating and differentiating cells and tissues especially in the brain. Iron deficiency in infancy has been associated with anemia and impaired neurodevelopmental outcomes that extend into childhood. Premature infants are at highest risk for iron deficiency because they are deprived of the iron accretion that occurs in the third trimester of pregnancy, are born with lower iron stores compared to their term counterparts, and have increased utilization and depletion of iron stores with their rapid growth rate.

In older populations, EOD iron supplementation is as effective as daily iron supplementation in the treatment of iron deficiency anemia, with studies revealing significantly fewer gastrointestinal side effects in those who are on EOD iron. Adults regulate their iron status through a feedback pathway involving hepcidin whereby iron-sufficient individuals will have upregulated hepcidin, which leads to decreased iron absorption and availability. Recent studies have revealed that pediatric patients and premature neonates regulate iron absorption through hepcidin in a similar fashion. Though the regulation of iron status through hepcidin has been studied in extremely premature neonates, the clinical effect of EOD dosing of iron has not yet been examined in this population.

This is a non-inferiority, blinded, randomized control trial designed to investigate if EOD iron is comparable to daily iron dosing in achieving iron replete status by reticulocyte hemoglobin measurements in premature infants.

ELIGIBILITY:
Inclusion Criteria:

* Children (Minor < 18 years of age)
* Neonates
* Hospitalized
* Premature infants who are on full enteral feeds and are started on oral iron
* Premature infants who completed 26 0/7 to 32 6/7 weeks' gestation at birth

Exclusion Criteria:

• Infants with known congenital anomalies or chromosomal abnormalities (such as Trisomy 18 or Trisomy 21), conditions that affect iron metabolism (such as thalassemia or hemochromatosis), bleeding disorders or coagulopathy, and received iron parenterally prior to randomization

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Determine if daily versus EOD oral iron at the same dose per kilogram per day will achieve similar incidence of iron replete status at 36 weeks PMA. | 1 Week-36 Weeks
  The iron replete status will be measured by reticulocyte hemoglobin (Ret-Hb) between EOD and daily iron supplementation.

SECONDARY OUTCOMES:
Characterize Ret-Hb levels in preterm infants. | 12-24 Months
  Laboratory data obtained from a query of the medical records will be used to characterize reticulocyte-hemoglobin (Ret-Hb) levels. The units used for Ret-Hb is "pg" or picograms.
Identify the number of blood transfusions received between enrollment and 36 weeks' PMA between two groups. | 12-24 Months
  Blood bank data obtained from a query of the medical records will be used to identify the number of blood transfusions received by each study participant.
Determine prevalence of bronchopulmonary dysplasia between two groups. | 12-24 Months
  A chart review of medical records will be used to identify which participants developed a diagnosis of bronchopulmonary dysplasia (BPD), clinically defined as the study participant requiring supplemental oxygen and/or respiratory support either at 28 days postnatal age or 36 weeks' postmenstrual age. The severity of BPD will be defined as that outlined by the 2019 Jensen guidelines.
Identify the number of subjects with sepsis between two groups. | 12-24 Months
  Microbiology data obtained from a query of medical records will be used to identify which participants developed blood, urine, or cerebrospinal fluid culture positive sepsis.
Identify the number with necrotizing enterocolitis (NEC)/gastrointestinal perforations between two groups. | 12-24 Months
  A chart review of medical records will be used to identify which participants developed necrotizing enterocolitis and/or gastrointestinal perforations.
Characterize growth between two groups. | 12-24 Months
  A query of medical records will be conducted to identify weight (grams), height (centimeters), and head circumference (centimeters) percentiles and velocity for the infants at birth up until 36 weeks' postmenstrual age.

CONTACTS AND LOCATIONS:
Overall Officials: Pratik K Parikh, MD, Principal Investigator — CHRISTUS Health; Richelle L Homo, MD, Principal Investigator — CHRISTUS Health; Brooke Army Medical Center
Locations (1):
- CHRISTUS Children's, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sriranjan J, Kalata C, Fusch G, Thomas K, Goswami I. Prevalence and Implications of Low Reticulocyte-Hemoglobin Levels among Extreme Preterm Neonates: A Single-Center Retrospective Study. Nutrients. 2022 Dec 16;14(24):5343. doi: 10.3390/nu14245343. PMID 36558502
- [Result] Wang Y, Wu Y, Li T, Wang X, Zhu C. Iron Metabolism and Brain Development in Premature Infants. Front Physiol. 2019 Apr 25;10:463. doi: 10.3389/fphys.2019.00463. eCollection 2019. PMID 31105583
- [Result] McCarthy EK, Dempsey EM, Kiely ME. Iron supplementation in preterm and low-birth-weight infants: a systematic review of intervention studies. Nutr Rev. 2019 Dec 1;77(12):865-877. doi: 10.1093/nutrit/nuz051. PMID 31532494
- [Result] Nii M, Okamoto T, Sugiyama T, Aoyama A, Nagaya K. Reticulocyte hemoglobin content changes after treatment of anemia of prematurity. Pediatr Int. 2022 Jan;64(1):e15330. doi: 10.1111/ped.15330. PMID 36321339
- [Result] Puia-Dumitrescu M, Tanaka DT, Spears TG, Daniel CJ, Kumar KR, Athavale K, Juul SE, Smith PB. Patterns of phlebotomy blood loss and transfusions in extremely low birth weight infants. J Perinatol. 2019 Dec;39(12):1670-1675. doi: 10.1038/s41372-019-0515-6. Epub 2019 Oct 3. PMID 31582812
- [Result] Bahr TM, Tan S, Smith E, Beauman SS, Schibler KR, Grisby CA, Lowe JR, Bell EF, Laptook AR, Shankaran S, Carlton DP, Rau C, Baserga MC, Flibotte J, Zaterka-Baxter K, Walsh MC, Das A, Christensen RD, Ohls RK; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Serum ferritin values in neonates <29 weeks' gestation are highly variable and do not correlate with reticulocyte hemoglobin content. J Perinatol. 2023 Nov;43(11):1368-1373. doi: 10.1038/s41372-023-01751-z. Epub 2023 Aug 18. PMID 37596391
- [Result] Karakoc G, Orgul G, Sahin D, Yucel A. Is every other day iron supplementation effective for the treatment of the iron deficiency anemia in pregnancy? J Matern Fetal Neonatal Med. 2022 Mar;35(5):832-836. doi: 10.1080/14767058.2021.1910666. Epub 2021 Apr 18. PMID 33866933
- [Result] Stoffel NU, Zeder C, Brittenham GM, Moretti D, Zimmermann MB. Iron absorption from supplements is greater with alternate day than with consecutive day dosing in iron-deficient anemic women. Haematologica. 2020 May;105(5):1232-1239. doi: 10.3324/haematol.2019.220830. Epub 2019 Aug 14. PMID 31413088
- [Result] von Siebenthal HK, Gessler S, Vallelian F, Steinwendner J, Kuenzi UM, Moretti D, Zimmermann MB, Stoffel NU. Alternate day versus consecutive day oral iron supplementation in iron-depleted women: a randomized double-blind placebo-controlled study. EClinicalMedicine. 2023 Nov 3;65:102286. doi: 10.1016/j.eclinm.2023.102286. eCollection 2023 Nov. PMID 38021373
- [Result] Pasupathy E, Kandasamy R, Thomas K, Basheer A. Alternate day versus daily oral iron for treatment of iron deficiency anemia: a randomized controlled trial. Sci Rep. 2023 Feb 1;13(1):1818. doi: 10.1038/s41598-023-29034-9. PMID 36725875
- [Result] German KR, Comstock BA, Parikh P, Whittington D, Mayock DE, Heagerty PJ, Bahr TM, Juul SE. Do Extremely Low Gestational Age Neonates Regulate Iron Absorption via Hepcidin? J Pediatr. 2022 Feb;241:62-67.e1. doi: 10.1016/j.jpeds.2021.09.059. Epub 2021 Oct 7. PMID 34626672
- [Result] Uyoga MA, Mikulic N, Paganini D, Mwasi E, Stoffel NU, Zeder C, Karanja S, Zimmermann MB. The effect of iron dosing schedules on plasma hepcidin and iron absorption in Kenyan infants. Am J Clin Nutr. 2020 Oct 1;112(4):1132-1141. doi: 10.1093/ajcn/nqaa174. PMID 32678434
- [Result] Manapurath RM, Gadapani Pathak B, Sinha B, Upadhyay RP, Choudhary TS, Chandola TR, Mazumdar S, Taneja S, Bhandari N, Chowdhury R. Enteral Iron Supplementation in Preterm or Low Birth Weight Infants: A Systematic Review and Meta-analysis. Pediatrics. 2022 Aug 1;150(Suppl 1):e2022057092I. doi: 10.1542/peds.2022-057092I. PMID 35921671
- [Result] MacQueen BC, Baer VL, Scott DM, Ling CY, O'Brien EA, Boyer C, Henry E, Fleming RE, Christensen RD. Iron Supplements for Infants at Risk for Iron Deficiency. Glob Pediatr Health. 2017 Apr 25;4:2333794X17703836. doi: 10.1177/2333794X17703836. eCollection 2017. PMID 28491927

DOCUMENTS (1):
  • Study Protocol (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT06555315/Prot_000.pdf